CLINICAL TRIAL: NCT05697731
Title: Evaluation of Vidiac Scores of Obese and Non-obese Patients Intubated by Videolaryngoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, aysun postaci, Ankara City Hospital, Ankara City Hospital Bilkent
Other Study IDs: E2-22-2939
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Vidiac Score; Videolaryngoscopy; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese: Vidiac score Mallampati score upper lip bite test Thyromental distance Mandible ramus length Mouth opening distance
  Interventions: Diagnostic Test: Vidiac Score
- non-obese: Vidiac score Mallampati score upper lip bite test Thyromental distance Mandible ramus length Mouth opening distance
  Interventions: Diagnostic Test: Vidiac Score

INTERVENTIONS:
Diagnostic Test: Vidiac Score — Vidiac score is a scoring system created according to the visibility of laryngeal structures under videolarnyngoscopy in patients with expected difficult intubation.

SUMMARY:
The aim of the study was to observe the vidiac score values of only patients with obesity as a risk factor for difficult intubation. Secondly, it was aimed to evaluate the number of intubation attempts and intubation time, vidiac scores between non-obese and obese patients and to reveal the differences, if any.

ELIGIBILITY:
Inclusion Criteria:

* All patients to be operated under general anesthesia and endotracheal intubation

Exclusion Criteria:

1. under 18 years old
2. The patient's refusal
3. Difficult airway story before
4. Congenital or previous airway anatomical disorder
5. Patients who have undergone airway surgery
6. Patients with a mass in the head and neck region

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients to be operated under general anesthesia and endotracheal intubation
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
vidiac score | during entubation
  Vidiac score is a scoring system created according to the visibility of laryngeal structures under videoingoscopy in patients with expected difficult intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Postacı, Assoc. Prof, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided